CLINICAL TRIAL: NCT04784026
Title: Comparison of Single and Dual Task Gait Performance in Pediatric Oncology Patients With Healthy Control Group
Brief Title: Dual Task Gait Performance in Pediatric Oncology Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2021/144
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Cancer
Keywords: pediatrics; neoplasms; gait
MeSH Terms: conditions — Neoplasms | interventions — Single Person

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control Group: Healthy children who come to Afyonkarahisar Ege Youth and Sports Club Association for the purpose of sports, newly registered and between the ages of 6-18 will constitute the control group of the study.
  Interventions: Other: Gait assessment (single); Other: Dual task gait assessment (motor+motor); Other: Dual tak gait assessment (motor+cognitive)
- Case Group: The sample of the study will be inpatient and outpatient pediatric patients between the ages of 6-18 who have been diagnosed with cancer in the Pediatric Hematology-Oncology Clinics of Afyonkarahisar Health Sciences University Health Application and Research Center Department of Pediatrics.
  Interventions: Other: Gait assessment (single); Other: Dual task gait assessment (motor+motor); Other: Dual tak gait assessment (motor+cognitive)

INTERVENTIONS:
Other: Gait assessment (single) — The single walk will be evaluated with a 10-meter walking test and a G-Walk portable device.
Other: Dual task gait assessment (motor+motor) — The dual task gait, 10-meter walking test and a motor (carrying a full water glass) will be combined with the task and evaluated with the G-Walk portable device.
Other: Dual tak gait assessment (motor+cognitive) — The dual task gait will be combined with a 10-meter walking test and a cognitive (1-back test) task and evaluated with the G-Walk portable device.

SUMMARY:
Cancer incidence, which is recognized as the leading cause of death in children worldwide, is gradually increasing.

Most studies on children who survive cancer show that the disease and its treatment have side effects and long-term late effects on the musculoskeletal system, physical function, gait and cognitive skills.

Therefore, dual task gait performance, in which cognitive and motor tasks are performed simultaneously, may be affected in pediatric oncology patients. The aim of this study is to compare gait performance in single and dual task conditions in pediatric oncology patients with healthy controls.

DETAILED DESCRIPTION:
Cancer incidence, which is recognized as the leading cause of death in children worldwide, is gradually increasing. About 300,000 children aged 0 to 19 are diagnosed with cancer each year, according to the international study where the International Agency for Research on Cancer collected data on neoplasms (malignant and non-malignant) diagnosed in individuals under 20 years of age between 2001-2010.

Most studies on children who survive cancer show that the disease and its treatment have side effects and long-term late effects on the musculoskeletal system, physical function, gait and cognitive skills. According to the study of Beulertz et al. (2016), active ankle dorsiflexion limitation, gait disturbances and decrease in walking efficiency were observed in all pediatric oncology patients, which have an important role in walking, not limited to children with bone tumors and central nervous system tumors.Intensive chemotherapy (eg methotrexate) and the use of radiation are thought to cause damage to cortical and subcortical white matter, resulting in late effects. Symptoms consistent with attention deficit disorder and mental processing speed, working memory, executive function and memory deficits put cancer survivors at an intellectual and academic disadvantage.

Therefore, dual task gait performance, in which cognitive and motor tasks are performed simultaneously, may be affected in pediatric oncology patients. The aim of this study is to compare gait performance in single and dual task conditions in pediatric oncology patients with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Healthy control group:

* Being in the age range of 6-18,
* To be physically, cognitively and mentally healthy,
* Open to communication enough to understand questions,
* Speaking and understanding Turkish,
* Approval has been obtained from the child and his / her family for the study and who agrees to participate in the study,

Case group:

* Able to walk alone without any walking aid,
* Open to communication enough to understand questions,
* Speaking and understanding Turkish,
* Approval has been obtained from the child and his / her family for the study and who agrees to participate in the study,
* Children between the ages of 6-18 will be included in the study

Exclusion Criteria:

Healthy control group:

* Any orthopedic or neurological impairment that would prevent walking;
* Having any mental disability that prevents cognitive task

Case group:

* Staying in an isolated room or having risk of infection (neutropenic, etc.),
* Any orthopedic or neurological impairment that could prevent walking;
* Having any mental disability that prevents cognitive task,
* Individuals with malignant hypertension or unstable heart disease (eg congestive heart failure) will not be included in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In this study, inpatient and outpatient children diagnosed with cancer in Afyonkarahisar Health Sciences University Health Application and Research Center Pediatric Hematology-Oncology Clinics will form the case group of the study.
  Healthy children who come to Afyonkarahisar Ege Youth and Sports Club Association to do sports and who have recently registered will form the control group of the research.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
gait speed | 20 minutes
  Gait speed is the time one takes to walk a specified distance on level surfaces over a short distance.
cadence | 20 minutes
  Cadence is the rate at which a person walk, expressed in steps per minute. The average cadence is 100 - 115 steps/min.
stride length | 20 minutes
  Stride length is defined as the distance between successive ground contacts of the same foot.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No